CLINICAL TRIAL: NCT01589185
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Assess the Safety, Pharmacokinetics, Efficacy and Pharmacodynamics of KBSA301 in Severe Pneumonia (S. Aureus)
Brief Title: Safety, Pharmacokinetics and Efficacy of KBSA301 in Severe Pneumonia (S. Aureus)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aridis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KBSA301-001
Record Dates: First submitted 2012-04-08; First posted 2012-05-01 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-03

CONDITIONS: Pneumonia Due to Staphylococcus Aureus
Keywords: Pneumonia; Monoclonal antibody; Staphylococcus aureus
MeSH Terms: conditions — Pneumonia; Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- KBSA301, a monoclonal antibody dose 1 (Experimental): 1 mg/kg KBSA301
  Interventions: Drug: KBSA301
- KBSA301, a monoclonal antibody dose 2 (Experimental): 3 mg/kg KBSA301
  Interventions: Drug: KBSA301
- KBSA301, a monoclonal antibody dose 3 (Experimental): 10 mg/kg KBSA301
  Interventions: Drug: KBSA301
- KBSA301, a monoclonal antibody dose 4 (Experimental): 20 mg/kg KBSA301
  Interventions: Drug: KBSA301
- Placebo (Experimental): KBSA301-placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KBSA301 — KBSA301 administered as a single intravenous infusion at dose 1, 2, 3 and 4.
  Other Names: AR301
  Arms: KBSA301, a monoclonal antibody dose 1; KBSA301, a monoclonal antibody dose 2; KBSA301, a monoclonal antibody dose 3; KBSA301, a monoclonal antibody dose 4
Drug: Placebo — Placebo administered as a single intravenous infusion
  Other Names: Placebo KBSA301
  Arms: Placebo

SUMMARY:
The objectives of this study are to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and clinical outcome of patients who have severe pneumonia caused by Staphylococcus aureus (S. aureus) after a single intravenous administration of KBSA301 in addition of standard of care antibiotic treatment.

DETAILED DESCRIPTION:
S. aureus is a leading cause of bloodstream, skin, soft tissue, and lower respiratory tract infections worldwide. The frequencies of both nosocomial and community-acquired S. aureus infections have increased steadily over the years and the treatment of these infections has become more challenging due to the emergence of multi-drug resistant strains (e.g. methicillin-resistant Staphylococcus aureus).

S. aureus has several virulence factors that contribute to the pathogenesis of the infection. Amongst them, alpha-toxin that is involved in the pathogenesis of pneumonia, as it leads to apoptosis and cell lysis, in particular lymphocytes, macrophages, alveolar epithelial cells, pulmonary endothelium, and thrombocytes.

In spite of preventive measures for S. aureus infections and current medical treatment (mostly antibiotic therapy, alone or in combination), there is a clear unmet medical need in the clinic for additional treatment options. Passive immunotherapy with monoclonal antibodies may improve treatment options for severe and life-threatening infections like those caused by S. aureus.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients ≥ 18 years and ≤ 70 years of age
* Severe pneumonia caused by S. aureus (either methicillin-resistant or methicillin-sensitive) managed in an ICU
* APACHE II of ≤30 at the time of diagnosis
* Identification of S. aureus
* Written informed consent provided by the patient, the relatives or the designated trusted person and/or according to local guidelines

Exclusion Criteria:

* Women of child bearing potential are excluded from the participation from the study unless they have a negative pregnancy test at baseline and during the course of the study. Postmenopausal women or females that have been surgically sterilized are allowed to participate.
* Hypersensitivity to excipients or to any prescribed medication
* Severe neutropenia, lymphoma or anticipated chemotherapy
* Patients who have long-term tracheostomy
* Current or recent investigational drug (within 30 days of enrollment, or 5 half-lives of the investigational compound, whichever is longer)
* Presence of meningitis, endocarditis, or osteomyelitis
* Acquired immune deficiency syndrome (AIDS) with cluster of differentiation 4 (CD4) count <200 cells/ml
* Known bronchial obstruction or a history of post-obstructive pneumonia.
* Active primary lung cancer or another malignancy metastatic to the lungs
* Cystic fibrosis, known or suspected Pneumocystis jiroveci pneumonia, or known or suspected active tuberculosis
* Immunosuppressive therapy
* Liver function deficiency
* Moribund clinical condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-05; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François M Laterre, MD, Principal Investigator — Université catholique de Louvain, Brussels, Belgium
Locations (18):
- United States (3):
  - Site 83, Jacksonville, Florida
  - Site 81, Oklahoma City, Oklahoma
  - Site 80, Houston, Texas
- Belgium (2):
  - Site 11, Brussels
  - Site 16, Liège
- France (11):
  - Site 41, Angers
  - Site 40, Angoulême
  - Site 32, Argenteuil
  - Site 34, Colombes
  - Site 36, Dijon
  - Site 35, La Roche-sur-Yon
  - Site 31, Limoges
  - Site 39, Lyon
  - Site 37, Nantes
  - Site 38, Orléans
  - Site 33, Tours
- Spain (2):
  - Site 51, Barcelona
  - Site 52, Barcelona

REFERENCES:
- [Result] Francois B, Mercier E, Gonzalez C, Asehnoune K, Nseir S, Fiancette M, Desachy A, Plantefeve G, Meziani F, de Lame PA, Laterre PF; MASTER 1 study group. Safety and tolerability of a single administration of AR-301, a human monoclonal antibody, in ICU patients with severe pneumonia caused by Staphylococcus aureus: first-in-human trial. Intensive Care Med. 2018 Nov;44(11):1787-1796. doi: 10.1007/s00134-018-5229-2. Epub 2018 Oct 21. PMID 30343314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment locations: Intensive Care Units. First subject enrolled: 16-May-2012. Last subject completed: 06-Sep-2016. The study was on administrative hold from 20-Nov-2012 to 24-Dec-2014.
Pre-assignment Details: Eligible patients were randomized based on evidence of severe pneumonia caused by S. aureus. All patients enrolled were intubated.
Period: Overall Study
Arm/Group | KBSA301, a Monoclonal Antibody Dose 1 | KBSA301, a Monoclonal Antibody Dose 2 | KBSA301, a Monoclonal Antibody Dose 3 | KBSA301, a Monoclonal Antibody Dose 4 | Placebo
Started | 6 | 8 | 10 | 8 | 16
Completed | 4 | 6 | 6 | 5 | 15
Not Completed | 2 | 2 | 4 | 3 | 1
Not completed — Death | 1 | 2 | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KBSA301, a Monoclonal Antibody Dose 1 | KBSA301, a Monoclonal Antibody Dose 2 | KBSA301, a Monoclonal Antibody Dose 3 | KBSA301, a Monoclonal Antibody Dose 4 | Placebo | Total
Number analyzed (Participants) | 6 | 8 | 10 | 8 | 16 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 5 | 4 | 12 | 31
  >=65 years | 3 | 1 | 5 | 4 | 4 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.97) | 49.1 (17.02) | 61.5 (10.30) | 60.6 (13.62) | 52.1 (16.23) | 56.6 (14.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 4 | 1 | 3 | 10
  Male | 4 | 8 | 6 | 7 | 13 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 8 | 9 | 8 | 15 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 0 | 1 | 0 | 0 | 1
  United States | 0 | 0 | 0 | 1 | 0 | 1
  France | 4 | 8 | 9 | 6 | 16 | 43
  Spain | 2 | 0 | 0 | 0 | 0 | 2
  United Kingdom | 0 | 0 | 0 | 1 | 0 | 1
Type of Pneumonia [Count of Participants; unit: Participants] — CABP = community-acquired bacterial pneumonia VABP = ventilator-acquired bacterial pneumonia HABP = hospital-acquired bacterial pneumonia
  Participants
    CABP | 1 | 3 | 0 | 1 | 4 | 9
    VABP | 5 | 4 | 7 | 5 | 5 | 26
    HABP | 0 | 1 | 3 | 2 | 7 | 13
Type of S. aureus Infection [Count of Participants; unit: Participants] — MRSA = methicillin-resistant S. aureus; MSSA = methicillin-susceptible S. aureus
  Participants
    MRSA | 2 | 0 | 0 | 2 | 2 | 6
    MSSA | 4 | 8 | 9 | 6 | 14 | 41
    Not confirmed | 0 | 0 | 1 | 0 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI = Body Mass Index measured in kg/m^2.
  kg/m^2 | 32.6 (9.14) | 28.1 (7.3) | 31.1 (6.15) | 29.1 (3.88) | 26.8 (5.39) | 29.0 (6.32)
Pa02/Fi02 Ratio [Mean (Standard Deviation); unit: ratio] — Ratio of arterial oxygen partial pressure (PaO2) to fractional inspired oxygen (FiO2).
  ratio | 146.7 (30.7) | 173.7 (38.36) | 138.8 (53.56) | 148.4 (34.49) | 140.7 (40.7) | 147.8 (41.32)
SOFA Score [Mean (Standard Deviation); unit: units on a scale (score)] — Sequential Organ Failure Assessment (SOFA) score. Improvement in the SOFA score is defined as a drop of at least one point from baseline to time of cure. SOFA points are given for increasing severity from 0 (least severe) to 4 (most severe) for each of six (6) physiological values. Total score is between 0 and 24. The mean of the computed SOFA score of all patients in a group is reported for each group.
  units on a scale (score) | 6.8 (1.64) | 8.8 (3.45) | 5.6 (1.51) | 6.8 (1.72) | 6.8 (2.86) | 6.9 (2.62)
APACHE II Score [Mean (Standard Deviation); unit: units on a scale (score)] — Acute Physiology and Chronic Health Evaluation (APACHE II) score. Improvement in the APACHE II score is defined as a drop of points from baseline to time of cure. APACHE II points are given for increasing severity calculated on twelve (12) physiological values for a total integer score from 0 to 71. The mean of the computed APACHE II score of all patients in a group is reported for each group.
  units on a scale (score) | 18.3 (3.01) | 21.5 (5.21) | 17.9 (4.15) | 19.5 (3.7) | 17.5 (4.9) | 18.7 (4.48)
CPIS Score [Mean (Standard Deviation); unit: units on a scale (score)] — The data refer to the modified Clinical Pulmonary Infection Score (CPIS) score. Improvement in the CPIS score is defined as a drop in points from baseline to time of cure. CPIS points are given for increasing severity from 0 (least severe) to 2 (most severe) for each of six physiological values. Total score is between 0 and 12. The mean of the computed CPIS score of all patients in a group is reported for each group.
  units on a scale (score) | 8.3 (1.63) | 9.6 (2.26) | 9.6 (2.26) | 9.6 (3.7) | 9.8 (1.28) | 9.6 (1.58)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Endpoint: All-Cause Mortality by Day 28
Description: A summary of the number (%) of patients who died on or before Day 28 (mITT population) is provided, by treatment group and overall.
Time Frame: At Day 28 post infusion (Day 0)
Population: The modified intent to treat (mITT) population corresponded to the safety (ITT) population minus one patient for which infection by S. aureus was not confirmed.
Measure: Count of Participants; unit: Participants
Groups:
- All Treatment Group: Sum of all four KBSA301 treatment groups (1 mg/kg, 3 mg/kg, 10 mg/kg and 20 mg/kg)
Arm/Group | KBSA301, a Monoclonal Antibody Dose 1 | KBSA301, a Monoclonal Antibody Dose 2 | KBSA301, a Monoclonal Antibody Dose 3 | KBSA301, a Monoclonal Antibody Dose 4 | Placebo | All Treatment Group
Number analyzed (Participants) | 6 | 8 | 9 | 8 | 16 | 31
Participants | 1 | 2 | 2 | 0 | 0 | 5

2. Secondary Outcome: Efficacy: All-Cause Mortality (End Of Study [EOS])
Description: A summary of the number (%) of patients who died on or before timepoints Day EOS (mITT population) is provided, by treatment group (overall) and placebo.
Time Frame: Patients who died during the specified timepoints (by EOS), up to day 107
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KBSA301, a Monoclonal Antibody Dose 1 | KBSA301, a Monoclonal Antibody Dose 2 | KBSA301, a Monoclonal Antibody Dose 3 | KBSA301, a Monoclonal Antibody Dose 4 | Placebo
Number analyzed (Participants) | 6 | 8 | 9 | 8 | 16
Participants
  Died on or before EOS | 1 | 2 | 2 | 0 | 1
  Survived on or before EOS | 5 | 6 | 7 | 8 | 15
Statistical Analysis 1: Comparison: KBSA301, a Monoclonal Antibody Dose 1 vs KBSA301, a Monoclonal Antibody Dose 2 vs KBSA301, a Monoclonal Antibody Dose 3 vs KBSA301, a Monoclonal Antibody Dose 4 vs Placebo; The number (%) of patients who died on or before end of study (EOS) was compared among all 5 groups. The mITT population was used; Test type: Superiority; p = 0.3962, Fisher Exact — < 0.1 is considered borderline significant

3. Secondary Outcome: Efficacy: All-Cause Mortality (Day 14)
Description: A summary of the number (%) of patients who died on or before timepoints Day 14 visit (mITT population) is provided, by treatment group (overall) and placebo.
Time Frame: Patients who died during the specified timepoints (Day 14)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KBSA301, a Monoclonal Antibody Dose 1 | KBSA301, a Monoclonal Antibody Dose 2 | KBSA301, a Monoclonal Antibody Dose 3 | KBSA301, a Monoclonal Antibody Dose 4 | Placebo
Number analyzed (Participants) | 6 | 8 | 9 | 8 | 16
Participants
  Died on or before Day 14 | 1 | 1 | 0 | 0 | 0
  Survived on or before Day 14 | 5 | 7 | 9 | 8 | 16

4. Secondary Outcome: Efficacy: All-Cause Mortality (Day 7)
Description: A summary of the number (%) of patients who died on or before timepoints Day 7 visit (mITT population) is provided, by treatment group (overall) and placebo.
Time Frame: Patients who died during the specified timepoints (Day 7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KBSA301, a Monoclonal Antibody Dose 1 | KBSA301, a Monoclonal Antibody Dose 2 | KBSA301, a Monoclonal Antibody Dose 3 | KBSA301, a Monoclonal Antibody Dose 4 | Placebo
Number analyzed (Participants) | 6 | 8 | 9 | 8 | 16
Participants
  Died on or before Day 7 | 0 | 1 | 0 | 0 | 0
  Survived on or before Day 7 | 6 | 7 | 9 | 8 | 16

5. Secondary Outcome: Efficacy: All-Cause Mortality (Day 21)
Description: A summary of the number (%) of patients who died on or before timepoints Day 21 visit (mITT population) is provided, by treatment group (overall) and placebo.
Time Frame: Patients who died during the specified timepoints (Day 21)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KBSA301, a Monoclonal Antibody Dose 1 | KBSA301, a Monoclonal Antibody Dose 2 | KBSA301, a Monoclonal Antibody Dose 3 | KBSA301, a Monoclonal Antibody Dose 4 | Placebo
Number analyzed (Participants) | 6 | 8 | 9 | 8 | 16
Participants
  Died on or before Day 21 | 1 | 2 | 1 | 0 | 0
  Survived on or before Day 21 | 5 | 6 | 8 | 8 | 16

ADVERSE EVENTS:
Time Frame: From time of treatment to day 107.
Description: Standard definitions were used.
Arm/Group | KBSA301, a Monoclonal Antibody Dose 1 | KBSA301, a Monoclonal Antibody Dose 2 | KBSA301, a Monoclonal Antibody Dose 3 | KBSA301, a Monoclonal Antibody Dose 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/6 | 2/8 | 2/10 | 0/8 | 1/16
Serious Adverse Events (participants affected / at risk) | 3/6 | 4/8 | 5/10 | 1/8 | 5/16
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 10/10 | 7/8 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KBSA301, a Monoclonal Antibody Dose 1 (N=6) | KBSA301, a Monoclonal Antibody Dose 2 (N=8) | KBSA301, a Monoclonal Antibody Dose 3 (N=10) | KBSA301, a Monoclonal Antibody Dose 4 (N=8) | Placebo (N=16)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Septic Shock (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KBSA301, a Monoclonal Antibody Dose 1 (N=6) | KBSA301, a Monoclonal Antibody Dose 2 (N=8) | KBSA301, a Monoclonal Antibody Dose 3 (N=10) | KBSA301, a Monoclonal Antibody Dose 4 (N=8) | Placebo (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Internal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site phlebitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acinetobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterobacter tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Severe acute respiratory syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 3 (3)
Wound abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrical burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (2)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 3 (3) | 3 (4) | 4 (4) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (1)
Carbon dioxide increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Prothrombin level abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral salt-wasting syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Quadriparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital lesion (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was not designed and not powered to demonstrate statistically significant differences between treatment groups. All efficacy results are descriptive and exploratory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days